CLINICAL TRIAL: NCT00542724
Title: An Open Label, Multi-Center, Randomized, Parallel Group Study Comparing the Efficacy and Safety of Insulin VIAject™ and Regular Human Insulin in Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biodel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIAject™-06J
Record Dates: First submitted 2007-10-05; First posted 2007-10-11 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Insulin; Diabetes Mellitus type I; Juvenile diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): VIAject™
  Interventions: Drug: VIAject™
- B (Active Comparator): Regular Human Insulin
  Interventions: Drug: Regular Human Insulin

INTERVENTIONS:
Drug: VIAject™ — Dosage as individually required
  Arms: A
Drug: Regular Human Insulin — Dosage as individually required
  Arms: B

SUMMARY:
The purpose of this study is to demonstrate equivalent blood glucose control in patients with type 1 diabetes mellitus with insulin VIAject™ and regular human insulin as prandial insulin and to demonstrate an equivalent safety profile for VIAject™ in comparison to regular human insulin.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients with type 1 diabetes must present with the following:

* Established diagnosis of type 1 diabetes for more than 1 year.
* HbA1c values of not more than 10.5%.
* Three months on a stable insulin regimen that meets the current standard of care and that includes at least two daily insulin injections.
* Age: 18 to 70 years.
* Body Mass Index: 18 - 38 Kg/m2.

Exclusion Criteria:

Patients presenting with any of the following will not be included in the study:

* Type 2 diabetes mellitus as determined by the investigator.
* History of frequent severe hypoglycemia within the prior six months.
* C-peptide > 1.0 ng/ml unless there is a documented history of ketoacidosis or a documented history of a positive anti GAD test.
* History of known hypersensitivity to any of the components in the study medication.
* History of severe or multiple allergies.
* Treatment with investigational diabetes drug in the last 3 months or treatment with any other investigational drug in the last 30 days before study entry.
* Current short-term treatment with systemic oral, injected, or inhaled corticosteroids. (inhaled corticosteroids may be allowed when the treatment is long-term).
* Progressive disease likely to prove fatal.
* History of malignancy within the past 5 years except for basal cell epithelioma.
* Known significant hepatic disease or serum AST or ALT values ≥ 3 X upper limit of normal or bilirubin levels ≥ 1.5 X upper limit of normal.
* Severe complications of diabetes mellitus including a history or finding of Stage III or IV diabetic retinopathy, proteinuria > 2+ by urine dipstick, serum creatinine of >1.8 mg/dl for males or >1.5 mg/dl for females, history of renal transplant, severe peripheral vascular disease which has resulted in an amputation, chronic foot ulcers claudication or absent pedal pulses.
* Known history of autonomic neuropathy.
* History of moderate to severe ketoacidosis within the 3 months preceding screening for the study.
* Current drug or alcohol abuse, or a history which in the opinion of the Investigator will impair patient safety or protocol compliance.
* Current significant cardiovascular, respiratory, gastrointestinal, hepatic, renal, neurological, psychiatric and/or hematological disease as evaluated by the Investigator.
* Blood donation within the last 30 days.
* A woman who is breast feeding.
* Pregnant women or women intending to become pregnant during the study.
* A sexually active woman of childbearing age not actively and consistently practicing birth control by using a medically accepted device or therapy.
* Abnormal ECG, safety lab or physical examination results which, in the opinion of the investigator, render the participation of the patient in the study to be inappropriate or unsafe.
* A history of lack of compliance with medical instructions, recent drug or alcohol abuse, or other reasons which, in the opinion of the investigator, render the participation of the patient in the study to be inappropriate or unsafe.
* Current significant diseases of the adrenal gland, pituitary gland or thyroid at the discretion of the investigator.
* Glomerular Filtration Rate < 40 ml/min.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2006-09; Primary Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 6 months
  To evaluate the mean changes in hemoglobin A1c (HbA1c) from baseline to the end of the study in subjects with type 1 diabetes after treatment for 6 months with Viaject in comparison to the mean changes in HbA1c from baseline to end of study in subjects treated with regular human insulin (RHI).

CONTACTS AND LOCATIONS:
Overall Officials: David C Klonoff, M.D., F.A.C.P., Principal Investigator — Diabetes Research Institute

REFERENCES:
- See also: Type 1 Diabetes study — http://www.biodel.com/